CLINICAL TRIAL: NCT01272700
Title: The Effect of Pressure Controlled Ventilation on the Pulmonary Mechanics in Prone Position Using the Wilson Frame: A Comparison With Volume Controlled Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2010-0201
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Herniation of Lumbar Vertebral Disc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCV (Experimental): Peak airway pressure were set to deliver a tidal volume of 10 ml/kg of ideal body weight
  Interventions: Procedure: volume control
- VCV (Active Comparator): After anesthetic induction, anesthesia maching were set to deliver a tidal volume of 10 ml/kg of ideal body weight
  Interventions: Procedure: pressure control

INTERVENTIONS:
Procedure: volume control — Volume controlled ventilation of tidal volume 10 ml/kg
  Arms: PCV
Procedure: pressure control — Pressure controlled ventilation for peak airway pressure to deliver tidal volume 10 ml/kg.
  Arms: VCV

SUMMARY:
Prone position in spinal surgery can increase airway pressure and decrease dynamic lung compliance by a frame used for postural stabilization. Also, it can increase hemodynamic instability such as reduced blood pressure by aggravating cardiac index.

Former study shows pressure controlled ventilation on the pulmonary mechanics can improve alveolar use and oxygenation than volume controlled ventilation. The latter one means controlling a patient's breathing completely through tidal volume and set breathing rate. This could be useful for the patients not possible to breath by themselves because it guarantees the perfect breathing.

The pressure controlled ventilation is used when there is a possibility to change a patient's environment. The pressure will be maintained steadily, but volume and flux will be changed. That means through the pressure already set, the whole breathing will be maintained from the beginning to end. If a patient's resistance is increased, the volume will be decreased even though the way of blood pressure control is same. However, the tidal volume per minute can be controlled somewhat and barotrauma can be decreased by controlling respiratory rate. Through this study, we are expecting the pressure controlled ventilation in prone position can improve lung mechanics and oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for lumbar spine surgery under general anaesthesia

Exclusion Criteria:

* Patients with coronary artery occlusive disease
* morbid obesity (body mass index ≥ 30 kg/m2)
* cerebrovascular disease and major obstructive or restrictive pulmonary disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
peak airway pressure | 30 minutes after prone position
  Record peak airway pressure on anesthesia mechanical ventilator after anesthesia induction and 30 minutes after prone positioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea